CLINICAL TRIAL: NCT04890119
Title: Prevalence Study of Amyloidosis in Patients With Surgery of Suspect Bilateral Carpal Tunnel (AMYLYONCARP)
Acronym: AMYLYONCARP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMYLYONCARP
Record Dates: First submitted 2021-05-06; First posted 2021-05-18 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Carpal Tunnel Syndrome Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: tenosynovial tissue biopsy — Biopsy of tenosynovial tissue during surgery for amyloid aggregate search

SUMMARY:
The purpose of this study is to evaluate the prevalence of amyloidosis in population of patient affected by suspect bilateral carpal tunnel with indication of surgery

ELIGIBILITY:
Inclusion Criteria:

* bilateral carpal tunnel with indication of surgery and judged suspect:
* age of 50 years old and more
* non-traumatic or undetermined neuropathic etiology or cardiac history (atrial arrhythmia or Heart Failure or cardiac stimulation) or family history of hereditary amyloidosis or monoclonal gammopathy

Exclusion Criteria:

* patient with diagnosis of amyloidosis
* traumatic bilateral carpal tunnel or linked to rheumatoid arthritis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of amyloid aggregate | During surgery
  Research of amyloid aggregate in tenosynovial tissue

SECONDARY OUTCOMES:
Typing of amyloid aggregate | During surgery
  Caracterization of amyloid aggregate in tenosynovial tissue

OTHER OUTCOMES:
Research of organ amyloidosis (context of standard care): exploratory | in the 3 months following surgery
  Among positive patients, additional exams will be performed in the context of standard care in order to research for organ amyloidosis: blood sampling, EKG, echocardiography and other organ exams according to type of amyloidosis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe SCHIELE, MD, Principal Investigator — Centre Hospitalier Saint Joseph Saint Luc
Locations (1):
- Centre Hospitalier Saint Joseph Saint Luc, Lyon, France

IPD SHARING:
Plan to Share IPD: No